CLINICAL TRIAL: NCT02257528
Title: A Phase II Evaluation of Nivolumab, a Fully Human Antibody Against PD-1, in the Treatment of Persistent or Recurrent Cervical Cancer
Brief Title: Nivolumab in Treating Patients With Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02021; NCI-2014-02021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PNRG-GY002_A01PAMDREVW01; NRG-GY002; NRG-GY002 (Other: NRG Oncology); NRG-GY002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Recurrent Cervical Carcinoma; Stage IV Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVB Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over approximately 60 minutes every 2 weeks for a maximum of 46 doses over 92 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies the side effects and how well nivolumab works in treating patients with cervical cancer that has grown, come back, or spread to other places in the body. Monoclonal antibodies, such as nivolumab, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the antitumor activity (proportion of objective response by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) of nivolumab with objective tumor response in patients with persistent, recurrent or metastatic carcinoma of the cervix.

II. To determine the nature and degree of toxicity of nivolumab as assessed by Common Terminology Criteria for Adverse Events (CTCAE) in patients with persistent, recurrent or metastatic carcinoma of the cervix.

SECONDARY OBJECTIVES:

I. To estimate the duration of progression-free survival (PFS) and overall survival (OS).

TERTIARY OBJECTIVES:

I. To systematically evaluate programmed cell death (PD)-1 and B7 homolog 1 (B7-H1) (i.e., PD-1 ligand) expression in tumor infiltrating lymphocytes (TILs) and cervical cancer cells and explore their correlations with objective response, PFS, and OS in nivolumab-treated patients with PD-1 and B7-H1 scoring results.

II. To explore the composition of immune infiltrates in tumor specimens/biopsies from primary and/or metastatic/recurrent sites with selected markers including (but not limited) to cluster of differentiation (CD)4+, CD8+, forkhead box P3 (FoxP3), CD25, lymphocyte activation gene-3 (LAG-3), T cell immunoglobulin mucin-3 (TIM-3), and inducible T-cell co-stimulator (ICOS) and their correlations to objective response, PFS and OS in nivolumab-treated patients.

III. To evaluate human papillomavirus (HPV) status and to explore the changes of pre- and post-immune therapy responses to HPV16/18/31/35/45 E7 antigens in patients peripheral blood lymphocytes (PBL) and serum using proliferative and interferon (IFN)-gamma enzyme-linked immunospot (ELISPOT) (cellular immunity) and serological (enzyme-linked immunosorbent assay [ELISA]) assays.

IV. To explore the levels of circulating tumor cells (CTCs) pre-treatment and at 8 and 12 weeks and their association with patient outcome.

OUTLINE:

Patients receive nivolumab intravenously (IV) over approximately 60 minutes every 2 weeks for a maximum of 46 doses over 92 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent, recurrent or metastatic squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix with documented disease progression (disease not amendable to curative therapy); NOTE: the following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric type adenocarcinoma, clear cell carcinoma and mesonephric carcinoma; histologic confirmation of the original primary tumor is required via the pathology report
* All patents must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target" lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Appropriate for study entry based on the following diagnostic workup:

  * History/physical examination within 28 days prior to registration
  * Imaging of target lesion(s) within 28 days prior to registration
  * Further protocol-specific assessments:

    * Recovery from adverse effects of recent surgery, radiotherapy or chemotherapy
    * Any other prior therapy directed at the malignant tumor including chemotherapy, biologic/targeted agents and immunologic agents must be discontinued at least three weeks prior to registration
    * Investigation agents must be discontinued for at least 30 days prior to registration
    * Any prior radiation therapy must be completed at least 4 weeks prior to registration
    * At least 4 weeks must have elapsed since any major surgery prior to registration
* Patients must have had one prior systemic chemotherapeutic regimen for management of persistent, recurrent or metastatic carcinoma of the cervix (e.g.; paclitaxel/cisplatin, paclitaxel/cisplatin/bevacizumab); chemotherapy administered concurrent with primary radiation (e.g.; weekly cisplatin) is not counted as a systemic chemotherapy regimen; adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is not counted as a systemic chemotherapy regimen (e.g.; paclitaxel and carboplatin for up to 4 cycles); NOTE: patients who have received more than one prior regimen are NOT eligible
* Performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/ul
* Platelets >= 100,000/ul
* Creatinine =< 1.5 x institutional upper limit of normal (ULN) or creatinine clearance (CrCl) >= 40 mL/min using Cockcroft-Gault formula
* Bilirubin =< 1.5 x ULN
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Normal thyroid function testing (thyroid stimulating hormone [TSH]) within 14 days prior to registration
* The patient or a legally authorized representative must provide study-specific informed consent authorization permitting release of personal health information prior to study entry

Exclusion Criteria:

* Patients who have had prior therapy with nivolumab or with an anti-PD-1, anti-PD-ligand (L)1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune check point pathways
* History of severe hypersensitivity reaction to any monoclonal antibody
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure and unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or nursing; women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug; WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IV/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab; women must not be breastfeeding

  * Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile or have undergone definitive radiation) do not require contraception
  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy of bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 month amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level greater than 40 mIU/mL
  * WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 23 weeks after the last dose of investigational product
  * Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform the treating physician immediately
* Patients with known brain metastases or leptomeningeal metastases are excluded unless the following conditions are met:

  * Metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete (must be confirmed within 28 days prior to the first dose of nivolumab administration)
  * There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

  * Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IRB), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patient with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

  * NOTE: patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, abdominal/pelvic fistula, gastrointestinal perforation, gastrointestinal (GI) obstruction and/or who require parenteral hydration and/or nutrition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D Santin, Principal Investigator — NRG Oncology
Locations (333):
- United States (333):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Santin AD, Deng W, Frumovitz M, Buza N, Bellone S, Huh W, Khleif S, Lankes HA, Ratner ES, O'Cearbhaill RE, Jazaeri AA, Birrer M. Phase II evaluation of nivolumab in the treatment of persistent or recurrent cervical cancer (NCT02257528/NRG-GY002). Gynecol Oncol. 2020 Apr;157(1):161-166. doi: 10.1016/j.ygyno.2019.12.034. Epub 2020 Jan 7. PMID 31924334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on 5/18/2015 and closed to accrual on 6/8/2016.
Groups:
- Treatment (Nivolumab): Patients were treated with 4 doses of IV nivolumab (3 mg/kg every 2 weeks), followed by an additional 42 doses 3 mg/kg every 2 weeks for a maximum of 46 doses until disease progression or adverse effects prohibit therapy.
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 26
Completed | 25
Not Completed | 1
Not completed — Never received study treatment | 1

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.6)
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 7
  40-49 years | 8
  50-59 years | 5
  60-69 years | 3
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response as Assessed by RECIST 1.1 Criteria
Description: Proportion of participants with objective tumor response. Objective tumor response is defined as complete or partial tumor response assessed by RECIST 1.1.
Time Frame: The average of study treatment time was 3.8 months.
Population: Eligible and evaluable participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 25
percentage of participants | 4 [0.9 to 100]

2. Primary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period as Assessed by CTCAE Version 4
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: Within 100 days of last protocol treatment
Population: Eligible and evaluable patients
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 25
participants
  Leukopenia | 1
  Thrombocytopenia | 1
  Neutropenia | 1
  Anemia | 3
  Other Investigations | 4
  Endocrine Disorders | 1
  Gastrointestinal disorders | 5
  General disorders & administration site conditions | 1
  Hepatobiliary disorders | 1
  Infections and Infestations | 1
  Metabolism and nutrition disorders | 5
  Musculoskeletal and connective tissue disorders | 1
  Neoplasms benign, malignant and unspecified | 2
  Other nervous system disorders | 1
  Reproductive system and breast disorders | 1
  Vascular disorders | 1

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. Progression is assessed by RECIST 1.1.
Time Frame: Time from study entry to time of progression or death, whichever occurs first, up to 5 years of follow-up.
Population: Eligible and Evaluable patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 25
months | 3.5 [1.9 to 5.1]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Time from study entry to time of death or the date of last contact, up to 5 years of follow-up
Population: Eligible and evaluable patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 25
months | 14.5 [8.3 to 26.8]

5. Other Pre Specified Outcome: Tumor Expressions of PD-1 and PD-L1 in Tumor Infiltrating Lymphocytes and Cervical Cancer Cells
Description: Spearman's correlation coefficient will be used to explore the associations of tumor expressions of PD-L1, PD-1 and other interested biomarkers with tumor response. Cox proportional hazards (PH) model will be utilized to evaluate the associations of these tumor expressions with PFS and OS. These expressions may also be dichotomized into high versus low values (cut at the median). Log-rank tests will be used to assess the associations of these dichotomized tumor expressions with PFS and OS. The corresponding hazard rations will be estimated by Cox PH models.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Immune Infiltration Related Biomarkers (i.e., CD4+, CD8+, FoxP3) in Tumor Specimens
Description: Immune infiltration related biomarkers (i.e., CD4+, CD8+, FoxP3) in tumor specimens will be associated with objective tumor response, PFS and OS in nivolumab-treated patients.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in the Immune Response to HPV 16/18/31/35/45 E7 Antigen in Peripheral Blood Lymphocytes and Serum
Description: Wilcoxon signed rank test (for interval or ordinal data) or McNemar's test (for binary data) may be utilized to examine whether the study treatment will change immune response to HPV 16/18/31/35/45 E7 antigen in peripheral blood lymphocytes and serum by changes in the measures of pre- and post-treatment immune response to HPV 16/18/31/35/45 E7.
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in the CTC Count
Description: Change in the CTC count and whether the CTC count is associated with objective response, PFS and OS in nivolumab-treated patients will be evaluated.
Time Frame: Baseline to up to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 5 years after are reported.
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 19/25
Serious Adverse Events (participants affected / at risk) | 12/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=25)
Hypothyroidism (Endocrine disorders) | 1
Colonic Obstruction (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Bile Duct Stenosis (Hepatobiliary disorders) | 1
Kidney Infection (Infections and infestations) | 1
Serum Amylase Increased (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab) (N=25)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 14
Palpitations (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Hyperthyroidism (Endocrine disorders) | 2
Endocrine Disorders - Other (Endocrine disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Colonic Obstruction (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 9
Bloating (Gastrointestinal disorders) | 1
Stomach Pain (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 11
Abdominal Distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 4
Pain (General disorders) | 2
Flu Like Symptoms (General disorders) | 1
Edema Limbs (General disorders) | 8
Fatigue (General disorders) | 15
Fever (General disorders) | 5
Chills (General disorders) | 2
Infusion Related Reaction (General disorders) | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 2
Vulval Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 1
Vaginal Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 3
Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Investigations - Other (Investigations) | 3
Weight Loss (Investigations) | 5
Serum Amylase Increased (Investigations) | 2
Platelet Count Decreased (Investigations) | 3
Lymphocyte Count Decreased (Investigations) | 3
Lipase Increased (Investigations) | 1
Creatinine Increased (Investigations) | 6
Neutrophil Count Decreased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 4
Alkaline Phosphatase Increased (Investigations) | 5
Alanine Aminotransferase Increased (Investigations) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 1
Recurrent Laryngeal Nerve Palsy (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 3
Urinary Urgency (Renal and urinary disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Fistula (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Cystitis Noninfective (Renal and urinary disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 2
Vaginal Hemorrhage (Reproductive system and breast disorders) | 3
Vaginal Fistula (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 3
Irregular Menstruation (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Thromboembolic Event (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT02257528/Prot_SAP_000.pdf